CLINICAL TRIAL: NCT06852027
Title: Evaluation of the Effects of Different Dietary Practices on Quality of Life and Eating Behavior in Children with Autism Spectrum Disorder
Brief Title: Different Dietary Practices in Children with Autism Spectrum Disorder
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Simge Gürel, Master student, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-15189967-050.04-593675
Record Dates: First submitted 2025-02-13; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Quality of Life; Eating Behavior; Autism Spectrum Disorder; gluten-free-casein-free diet; feingold diet
MeSH Terms: conditions — Autism Spectrum Disorder; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gluten-Free-Casein-Free Diet (Experimental): The Gluten-free Casein-free diet is one of the most researched diets for Autism Spectrum Disorder. This diet is based on the elimination of foods containing gluten and casein. In this arm, children between the ages of 3 and 10 will be subjected to a Gluten-free-Casein-free diet for 12 weeks. Children will be controlled for compliance with the diet every two weeks.
  Interventions: Other: Different Dietary Practices
- Feingold Diet (Experimental): The Feingold Diet was originally developed for Attention Deficit and Hyperactivity Disorder, it is thought to be effective in symptomatic treatment due to enzyme deficiency in children with Autism Spectrum Disorder, but there are not enough studies on it. The Feingold Diet is one of the most researched diets for Autism Spectrum Disorder. This diet is based on the elimination of foods containing gluten and casein. In this arm, children between the ages of 3 and 10 will be subjected to a the Feingold Diet diet for 12 weeks. Children will be controlled for compliance with the diet every two weeks.
  Interventions: Other: Different Dietary Practices
- Control (No Intervention): the arm receives no intervention during the study. (CONTROL GROUP). Children in this group will be monitored every 2 weeks for 12 weeks.

INTERVENTIONS:
Other: Different Dietary Practices — The aim was to investigate the effects of Gluten-Casein-Free Diet and Feingold Diet on gastrointestinal complaints in children with Autism Spectrum Disorder.
  Arms: Feingold Diet; Gluten-Free-Casein-Free Diet

SUMMARY:
The aim of this study is to investigate the effects of gluten-free casein-free diet and feingold diet on gastrointestinal system (GI) symptoms , eating behavior and quality of life in children with autism spectrum disorder. Research questions are below:

Is there a difference in the effects of a gluten-free-casein-free diet and the Feingold Diet on GI symptoms? Is there a difference in the effects of a gluten-free-casein-free diet and the Feingold Diet on eating behavior? Is there a difference in the effects of a gluten-free-casein-free diet and the Feingold Diet on quality of life?

DETAILED DESCRIPTION:
Autism Spectrum Disorder is defined as different neurodevelopmental disorders characterized by social communication, restrictive, repetitive, and typical behaviors and interests. Although it is not known precisely how the disease develops, literature reviews see genetic and environmental factors as the leading causes. The prevalence of Autism Spectrum Disorder is increasing day by day. There is no treatment for Autism Spectrum Disorder in light of the latest data. The applications made are primarily aimed at reducing stereotypical behaviors. Children with Autism Spectrum Disorder often experience gastrointestinal complaints such as diarrhea, constipation, abdominal pain, bloating, and gas. In addition, children with ASD also experience food selectivity, restrictive/avoidant feeding disorder, food neophobia, and nutritional problems due to sensory sensitivity. Considering these conditions, it is thought that dietary therapy may also be effective in the symptomatic treatment of Autism Spectrum Disorder with the support of studies conducted in recent years.

The Gluten-free Casein-free diet developed for Autism Spectrum Disorder is among the most researched diets. This diet is based on the elimination of foods containing gluten and casein. Although the other diet discussed in this study, the Feingold Diet, was developed initially for Attention Deficit and Hyperactivity Disorder, it is thought that it may be effective in symptomatic treatment due to enzyme deficiency in children with ASD. However, there are not enough studies on it. This study aimed to examine the effects of the Gluten-Casein-Free Diet and the Feingold Diet on gastrointestinal complaints in children with Autism Spectrum Disorder using the Scale of Eating Time Behaviors in Children with Autism (BAMBI), the Gastrointestinal Sensitivity Index and the Quality of Life Scale for Children. The study was planned to be conducted with 45 children with ASD between the ages of 3-10 registered at the Efeler Autism Life Center affiliated with the Efeler District Municipality of Aydın Province. Therefore, the necessary permissions will be obtained from the Efeler Autism Life Center, and the study will be submitted to the ethics committee for approval. The research data will be analyzed using the SPSS 22 (Statistical Package for the Social Sciences) program. Numbers and percentage distributions for descriptive feature data; correlation analyses will be used to determine the relationship and analyses appropriate for nonparametric and parametric data between the data.

ELIGIBILITY:
Inclusion Criteria:Children with autism between the ages of 3-10 registered at Efeler Autism Life Center in Aydın province.

The criteria for inclusion for the gluten-free-casein-free diet are as follows:

* Not having diseases such as celiac, lactose intolerance
* Not having previously applied a gluten-free diet, gluten-free casein-free diet, lactose-free diet
* Having gastrointestinal complaints

The criteria for inclusion for the Feingold Diet are as follows:

* Not having been diagnosed with attention deficit and hyperactivity disorder
* Not having previously taken the Feingold diet
* Not having any food allergies

Exclusion Criteria:People who do not comply with the diet or do not respond to the survey will be excluded from the study and the information obtained will not be used for the research.

* The patient is breastfed
* The patient has any chronic disease
* The patient has any psychiatric disease

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | Baseline and 3 months
  It will be evaluated whether there is a difference in the effects of the gluten-free-casein-free diet and the Feingold Diet on the gastrointestinal system. The evaluation will be made using the Gastrointestinal Sensitivity Index.
  Gastrointestinal Sensitivity Index: The GI sensitivity index assesses 0-17 points. A score of seven and above is a severe symptom in the child. The Gastrointestinal Sensitivity Index is applied by hospital personnel. It was prepared to examine children's digestive problems and their changes according to periods. The test consists of nine headings under the heading of symptoms: "Constipation, Diarrhea, Average Stool Density, Abdominal Hardness, Stool Odor, Flatulence, Abdominal Pain, Unexplained Daytime Irritability, Nighttime Awakening, and Abdominal Hardness." Each heading was matched with the answers numbered "0, 1, 2" and the sensitivity index was obtained.
Eating behaviors | Baseline and 3 months
  It will examine whether there is a difference between the effects of the gluten-free-casein-free diet and the Feingold Diet on eating behavior.
  Brief Autism Mealtime Behaviors Inventory (BAMBI): It was adapted into Turkish by Meral and Fidan in 2014. The scale consists of 18 items. It consists of three subscales: limited food variety, refusal, and autism-related behavioral characteristics. Items 3, 9, 10, and 15 are reverse-scored. Each item is scored as 1 for never, 2 for rarely/rarely, 3 for occasionally/sometimes, 4 for often, and 5 for always, according to its frequency of occurrence. The BAMBI-total score and subscale scores are as follows: For the limited food variety score, the total score of items 10, 11, 13, 14, 15, 16, 17, and 18 is evaluated; for the food refusal score, the total score of items 1, 2, 4, 7 and 8 is evaluated; and for the autism-specific behavior score, the total score of items 3, 5, 6, 9 and 12 is evaluated. High scores from the total and subscales indicate
Pediatric Quality of Life | Baseline and 3 months
  It will examine whether there is a difference between the effects of the gluten-free-casein-free diet and the Feingold Diet on quality of life.
  The Pediatric Quality of Life Inventory (PedsQL): The Children's Quality of Life Questionnaire (PedsQL) was developed by Varni and colleagues in 1999 to assess the health-related quality of life of children and adolescents between the ages of 2 and 18. The scale has four separate forms organized according to age group characteristics for the 2-4, 5-7, 8-12, and 13-18 age groups. The Turkish validity and reliability studies of the forms for the 5-7 age group were conducted by Üneri et al., and the Turkish validity and reliability studies of the forms for the 8-12 and 13-18 age groups were conducted by Memik et al. The scale, which has a parent-only form for the 2-4 age group, has both parent and child forms for other age groups. The scale has four subscales that question physical, emotional, social, and school-related functionality. While a fi

CONTACTS AND LOCATIONS:
Locations (1):
- Aydin province Efeler Autism Life Center, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No